CLINICAL TRIAL: NCT01427244
Title: A Phase II Evaluation of Trastuzumab In Patients With HER2 Positive Persistent Or Recurrent Vulvar Paget's Disease
Brief Title: Evaluation of Trastuzumab In Patients With HER2 Positive Persistent Or Recurrent Vulvar Paget's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1004006704
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Paget's Disease of the Vulva
Keywords: HER2+; Histologic confirmation; measurable disease; HER2 positive; HER2 overexpression; persistent vulvar Paget's disease; recurrent vulvar Paget's disease
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab (Experimental): Open Label
  Interventions: Drug: trastuzumab

INTERVENTIONS:
Drug: trastuzumab — monoclonal antibody

SUMMARY:
This is a phase II open-label study of the activity and safety of trastuzumab in patients with vulvar Paget's disease with overexpression of HER2 on biopsy.

DETAILED DESCRIPTION:
The primary objective will be to estimate the anti-tumor activity of trastuzumab by evaluating the response to trastuzumab therapy in patients with recurrent or persistent vulvar Paget's disease demonstrating HER2/neu overexpression by immunohistochemistry and/ or FISH ((fluorescence in situ hybridization).

The secondary objectives:

* To evaluate the quality of life, based on the severity of the patients' vulvar itching on a 4-point verbal rating scale from 0 to 3 (0=no itching, 1=mild itching/ bothersome, 2=moderate itching/ troublesome, 3=severe itching/ extremely troublesome) as well as on the severity of the patients' vulvar pain on a numeric pain scale from 0-10 (0=no pain, 1-3=mild pain, 4-6=moderate pain, 7-10=severe pain).
* To assess the frequency and severity of observed adverse effects
* To assess the frequency/ incidence of HER2 in Paget's disease of the vulva

ELIGIBILITY:
Inclusion Criteria:

* recurrent or persistent vulvar Paget's disease with overexpression of HER2 by immunohistochemistry and or fluorescence in situ hybridization (FISH)
* Biopsy for histologic confirmation
* Measurable disease
* Karnofsky score of 50-100
* recovered from effects of recent surgery, radiotherapy, or chemotherapy
* free of active infection requiring antibiotics
* adequate bone marrow function,renal function,hepatic function,cardiac function,WOCBP-neg.serum pregnancy,meet requirements in section 7.0

Exclusion Criteria:

* no measurable disease
* tumors not HER2 positive by immunohistochemistry FISH
* prior therapy with any anti-HER2 monoclonal antibody preparation
* Karnofsky score of 0-40
* other invasive malignancies, with the exception of non-melanoma skin cancer
* Patients requiring supplemental oxygen
* unstable medical conditions in the opinion of the treating physician place them at unacceptably increased risk from trastuzumab therapy
* Patients with active or unstable cardiac disease, or myocardial infarction within 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
measurement of the longest diameter for all target lesions | 5 years
  Where possible measurement of the target lesion size in 2 perpendicular diameters will be required for follow up. A Change in the product of these 2 diameters affords some estimate of change in tumor size and hence therapeutic efficacy. Response criteria will be based on the RECIST modified response evaluation criteria (appendix I).The reporting of these changes will be on an individual case basis and will be in terms of the best response achieved by that case.

SECONDARY OUTCOMES:
To assess the safety profile of trastuzumab in persistent or recurrent vulvar Paget's disease | 5 years
  To assess the safety profile for all patients who receive any amount of trastuzumab will be evaluable for toxicity.At each visit, a brief focused history will be obtained and any indication of treatment related toxicity will be evaluated by appropriate examination and/or laboratory/radiographic studies using the CTCAE v4.0 toxicity grades for both laboratory and non-laboratory data.The evaluation period should extend from date of first treatment until 30 days (or longer if so specified) from the last dose, or until resolution from all acute toxicities associated with the drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Rutherford, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut, United States